CLINICAL TRIAL: NCT05756270
Title: Clinical Applicability of Pseudo-continuous Arterial Spin Labeling as a Substitute for FDG-position Emission Tomography in MCI and SCD Patients
Brief Title: Clinical Applicability of pCASL as a Substitute for FDG-PET in MCI and SCD Patients
Acronym: CAPE
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: CAPE
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Mild Cognitive Impairment; Subjective Cognitive Decline
Keywords: pseudo-continuous arterial spin labeling; fluorodeoxyglucose positron emission tomography; mild cognitive impairment; biomarkers; subjective cognitive decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and CSF samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: pCASL — Brain 3 Tesla MRI with pCASL sequence

SUMMARY:
The goal of this observational study is to compare cerebral perfusion patterns with pseudo-continuous arterial spin labeling (pCASL) and brain metabolism patterns with fluorodeoxyglucose-position emission tomography (FDG-PET) in patients with mild cognitive impairment (MCI) and subjective cognitive decline (SCD). The main questions it aims to answer are:

* Do pCASL sequences identify hypoperfusion patterns that correlate well with FDG-PET hypometabolic patterns?
* Are there differences in this correlation in terms of cerebrospinal fluid (CSF) profiles?
* Can hypoperfusion patterns in pCASL predict conversion to dementia? Participants will undergo brain 3 Tesla magnetic resonance imaging (MRI), FDG-PET, lumbal puncture and blood collection to analyze amyloid beta and tau, yearly detailed neuropsychological tests for three years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild cognitive impairment or subjective cognitive decline according to established criteria
* Clinical Dementia Rating scale of 0 or 0.5
* Signed informed consent before study entry

Exclusion Criteria:

* Contraindication to brain MRI, FDG-PET or lumbar puncture
* Secondary causes of cognitive decline
* Known major neurological or psychiatric comorbidities
* History of substance or alcohol abuse
* Known causes of cerebral brain perfusion alterations
* Enrollment in anti-amyloid or anti-tau drugs trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mild cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between brain hypoperfusion and brain hypometabolism at baseline | Baseline
  The investigators will correlate cerebral perfusion indices and standardized uptake value ratios (SUVr) ratios for each pre-specified region of interest (ROI) within statistical parametric mapping (SPM) Automatic Anatomic Labeling (AAL), after coregistration on T1 sequences
Correlation between brain hypoperfusion and brain hypometabolism at baseline according to CSF profile | Baseline
  The investigators will correlate cerebral perfusion indices and SUVr for each pre-specified ROI (region of interest) within SPM Automatic Anatomic Labeling (AAL), after coregistration on T1 sequences. This analysis will be done within subgroups according to CSF status according to amyloid beta, phosphorylated tau and total tau.

SECONDARY OUTCOMES:
Differences among brain hypoperfusion patterns according to amyloid and tau status | Baseline
  The investigators will analyze differences in brain perfusion indices for each ROI among patients wit amyloid positive status, amyloid and tau negative status, and amyloid negative - tau positive status
Correlations between brain hypoperfusion and neuropsychological tests | Baseline, 1 year, 2 years
  The investigators will perform correlations between brain hypoperfusion indices for each ROI and various neuropsychological (NPS) test scores
Predictive properties of brain hypoperfusion and brain hypometabolism for conversion to dementia | 1 year, 2 years
  The investigators will analyze correlations between each ROI hypoperfusion and conversion to dementia rates within the prespecified time frame. In case of significant associations, a receiver operating characteristic curve (ROC) analysis will be carried out to individuate optimal cut-offs for cerebral blood flow indices and SUVr to predict conversion of dementia
Correlations between brain hypoperfusion and CSF and blood biomarkers | Baseline
  The investigators will perform correlations between brain hypoperfusion indices for each ROI and values of CSF and blood amyloid beta, phosphorylated tau and total tau

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS San Gerardo dei Tintori, Monza, MB, Italy